CLINICAL TRIAL: NCT02739074
Title: Effectiveness of Metal Protheses Covered in "Diabolo" in Treatment of Necrosis of Origin Pancreatic: Trial "DIABOLOPIG"
Acronym: DIABOLOPIG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 15-PP-01
Record Dates: First submitted 2016-03-31; First posted 2016-04-14 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2016-03

CONDITIONS: Pancreatic Diseases
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Endoscopic treatment of pancreatic necrosis complicated by trans digestive track (duodenal or gastric) has become a standard technique validated. The rate of high technical and clinical success (76 to 91% in 3 months) and the lower morbidity in the literature explains that validation. However this treatment is done at the cost of a higher median number of treatment sessions (4-5) explaining prolonged hospitalization, delays in rehabilitation and potentially high costs. The constant improvement of therapeutic endoscopy equipment was allowed to see the advent of metal prosthesis completely covered by a membrane allowing them endoscopic extraction with ease. It has thus been recently developed short prostheses, of large diameter (up to 15/16 mm), with broad flange (or stent "diabolo") to be considered for use in the drainage of digestive peri collections. Few studies respectively determined the effectiveness of this type of prosthesis in the drainage of peri digestive collections Under echo endoscopy and treatment of necrosis of pancreatic origin. The purpose of this work is to evaluate multicenter prospective clinical and technical efficiency of laying completely covered stent "diabolo" in echo endoscopy for the treatment of necrosis of pancreatic origin.

ELIGIBILITY:
Inclusion Criteria:

Presence of peri gastric or duodenal collection type WOPN to imaging according to the Atlanta criteria (Banks Gut 2013) with predominantly solid component (> 50%) for imaging, requiring necrosectomy for:

* Pain and / or,
* necrosis infection (positive necrosis culture, gas bubble presence in the collection on imaging, persistent sepsis or deterioration of the patient's condition despite optimal reanimation support without documented infection) and / or,
* High Occlusion (vomiting, food intolerance and gastric stasis at imaging)

Exclusion Criteria:

* Severe coagulation disorders or hemostasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment is in hospital, all patients being hospitalized in case of complicated pancreatic necrosis requiring treatment. The treatment will be done like habitually by using a Diabolo prothesis. Investigators physicians will all doctors gastro enterology experts in interventional endoscopy supports daily basis patients with acute pancreatitis. Further investigation centers are tertiary referral centers authorized to support acute complicated pancreatitis.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Rate of patients who complete treatment of pancreatic necrosis | 3 months
  Rate of patients who complete treatment of pancreatic necrosis was obtained (> 80% and amendment of symptoms) after a single necrosectomy endoscopic session with a covered metal prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy VANBIERVLIET, Dr, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France